CLINICAL TRIAL: NCT06722170
Title: A Study on the Safety, Tolerability, and Preliminary Efficacy of EH002 in the Treatment of DFNB9 Congenital Deafness
Brief Title: A Study of EH002 Gene Therapy for Otoferlin Gene Mutation-mediated Hearing Loss
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yilai Shu (Other)
Responsible Party: Sponsor-Investigator, Yilai Shu, Director, Principal Investigator, Clinical Professor, Eye & ENT Hospital of Fudan University
Organization: Eye & ENT Hospital of Fudan University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2024199
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: DFNB9; Congenital Hearing Loss; Hearing Loss, Sensorineural
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dose escalation: 50-μl dose group (Experimental)
  Interventions: Genetic: EH002 administration
- Dose escalation: 100-μl dose group (Experimental)
  Interventions: Genetic: EH002 administration
- Dose escalation: 150-μl dose group (Experimental)
  Interventions: Genetic: EH002 administration
- Dose escalation: 25-μl dose group (Experimental)
  Interventions: Genetic: EH002 administration

INTERVENTIONS:
Genetic: EH002 administration — EH002 was administered into one or both ears via intracochlear injection.

SUMMARY:
The study is designed to evaluate the safety, tolerability, and preliminary efficacy of EH002 for the treatment of congenital deafness caused by mutations in the OTOF gene. Participants may receive one or two injections of the EH002 gene therapy in one or both ears.

ELIGIBILITY:
Inclusion Criteria:

1. The participant and/or their legal guardian must provide informed consent before the study, voluntarily sign the written informed consent form, and be willing to attend follow-up visits as scheduled by the study.
2. The participant must communicate effectively with the investigator and comply with the investigator's requirements, with the assistance of a legal guardian if necessary. Young children without mature language skills must be able to cooperate and comply with the investigator's requirements with the help of a legal guardian.
3. The participant and/or legal guardian must understand the study correctly and have appropriate expectations regarding the potential benefits.
4. The participant must be at least 6 months old, with no restrictions on gender.
5. The participant must be diagnosed with DFNB9 congenital deafness, confirmed by genetic testing showing homozygous or compound heterozygous mutations in the OTOF gene.
6. Audiological inclusion criteria: Severe or profound hearing loss (≥65 dB).
7. The participant must meet the surgical requirements, including the absence of middle- or inner-ear malformations, vestibulocochlear nerve developmental abnormalities, and ear inflammation, as confirmed by CT or MRI scans within 3 months or at the time of screening. Additionally, the participant must be deemed eligible for surgery.

Exclusion Criteria:

1. The genetic diagnosis does not indicate an OTOF mutation.
2. Other types of deafness that are unsuitable for otological surgery, such as middle- or inner-ear developmental abnormalities or malformations, vestibulocochlear nerve abnormalities, conductive hearing loss, mixed hearing loss, or malformation syndromes, as detected by CT or MRI scans within 3 months.
3. Pre-existing otological conditions that would interfere with the planned surgery or the interpretation of study endpoints, such as acute or chronic otitis media, Meniere's disease, acoustic neuroma, or unrecovered sudden sensorineural hearing loss.
4. A history of substance abuse, or treatment with any known ototoxic drugs (e.g., aminoglycosides, cisplatin, loop diuretics) within the last 6 months, or antiviral medications or immunotherapy within the last 3 months, or vaccination within the last month.
5. Individuals with compromised immunity or a history of immunodeficiency, including HIV-positive status, other acquired or congenital immunodeficiency disorders, or a history of organ transplantation.
6. Patients with severe systemic diseases or severe acute illnesses, such as tuberculosis, active hepatitis B or C infection, active herpes zoster infection, pancreatitis, renal insufficiency, or gastrointestinal ulcers.
7. Patients with surgical or anesthetic contraindications as determined by the surgeon, anesthesiologist, or designated personnel. This includes those who have had a cardiovascular or cerebrovascular event within the last 6 months, such as myocardial infarction, heart failure, angina, stroke, transient ischemic attack, or any other cardiac condition deemed unsuitable by the investigator or an allergy to any planned medications.
8. Currently participating in or planning to participate in any interventional clinical trial involving drugs or devices within the next year or having received the last dose of another clinical trial within 5 half-lives.
9. Presence of an implant in the ear (on the side intended for surgery) at the time of screening, such as a cochlear implant.
10. Neutralizing antibody titer against AAV1 >1:2000.
11. Presence of other severe congenital disorders.
12. A history of definite neurological or psychiatric disorders, including epilepsy or dementia.
13. Patients requiring long-term anticoagulant therapy that cannot be temporarily discontinued.
14. A history of chemotherapy or radiation therapy.
15. Any other condition that, in the opinion of the investigator, makes the participant unsuitable for this clinical study.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
The incidence of dose-limited toxicity and the incidence of serious adverse events or adverse events | 26 weeks

SECONDARY OUTCOMES:
Changes in hearing level relative to baseline level | 26 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No